CLINICAL TRIAL: NCT06702293
Title: Development and Testing of a Digital Psychological Tool to Improve Symptom Burden in Dermatology Patients
Brief Title: Use of a Digital Psychotherapeutic App to Reduce Symptom Burden in Dermatology Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Skin Centre, Singapore (Other); National University of Singapore (Other); KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022/00751
Record Dates: First submitted 2024-10-10; First posted 2024-11-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-09

CONDITIONS: Eczema; Psoriasis; Urticaria
Keywords: digital health; eczema; psoriasis; urticaria; healthservices research; digital; mental health
MeSH Terms: conditions — Eczema; Psoriasis; Urticaria; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): This fully automated and self-administered intervention will be delivered via a Health Insurance Portability and Accountability Act (HIPAA) compliant mobile app developed in collaboration with Intellect Inc., a Singapore-based mobile health company with broad reach and prior research collaborations in the Asia Pacific region. A detailed discussion focusing on the engineering of the application including the user interface, data acquisition and curation technology, security and privacy assurance is available from the authors.
  Interventions: Behavioral: Digital psychotherapeutic intervention
- Control (Active Comparator): Participants in the active control group will download use the Healthy365 app, a mobile health application managed by the Singapore government's Health Promotion Board. The Healthy365 app offers a variety of useful general health-related content which are not specific to skin disease. These include personalized health tracking, participation in fitness challenges, access to nutritional guidance, and personalized lifestyle recommendations.
  Interventions: Behavioral: Healthy365

INTERVENTIONS:
Behavioral: Digital psychotherapeutic intervention — Mobile app comprising various psychobehavioural tools to educate, enhance self-efficacy and coping and promote wellness in dermatological patients.
  Other Names: mobile app
  Arms: Intervention Arm
Behavioral: Healthy365 — Mobile application by the Health Promotion Board (HPB) Singapore which aims to encourage users to adopt a healthier lifestyle.
  Arms: Control

SUMMARY:
Skin diseases, despite low mortality, significantly impair quality of life. This randomised controlled trial evaluates the efficacy of a digital toolkit comprising psychotherapeutic strategies in reducing QoL burden in patients with chronic inflammatory skin conditions. This toolkit is hosted on a mobile application and will be used by study participants randomised to the intervention arm over the 32 week study period.

DETAILED DESCRIPTION:
Chronic inflammatory skin diseases, despite low mortality, significantly impair quality of life. Up to 80% of dermatological patients experience severe itch and poor sleep, and related such mental health challenges as anxiety and depression. The relationship between skin diseases and mental health highlights the challenges that doctors face in treating these conditions. Existing psychotherapeutics such as Mindfulness training, Cognitive Behavioural Therapy, and Acceptance and Commitment Therapy are widely used and effective in the treatment of mental health illness. However, there is limited evidence on the application of such interventions in dermatology and most mental health apps lack robust clinical evaluation. We report the design of a randomised controlled trial to evaluate the efficacy and implementation of a mobile app containing dermatology-specified psychotherapeutic strategies in reducing QoL burden.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis, eczema or chronic urticaria diagnosed by a dermatologist
* Aged 16 or older
* Peak pruritus intensity of 4 or more on a 11-point numerical rating scale (0-10, with 10 representing worst itch)
* Able to engage with a mobile application in the English language

Exclusion Criteria:

* Patients with active psychiatric symptoms (e.g. active suicidal ideation, psychosis, delusions)
* Patients with unstable psychiatric condition, characterized by

  o Hospital inpatient admission for a psychiatric condition or initiation of a psychotropic medication in the prior 3 months
* Patients with unstable dermatological condition, characterized by

  * Recent flare of the skin condition within the last 2 weeks, including diagnosis of a flare by a doctor, use of systemic steroids, oral antibiotics, wet wrap rescue therapy, oral antivirals, or increase in frequency of phototherapy or dose of systemic medications for the dermatological condition within the last 2 weeks OR
  * Any of the following within 3 months

    * inpatient admission for a dermatological condition
    * Initiation of phototherapy
    * Initiation of systemic therapy (conventional immunosuppressive agent, biologics, JAK inhibitors) within the last 3 months.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Skin-specific quality of life impairment | baseline, week 8
  Dermatology Life Quality Index (DLQI). Minimum Score: 0 (no impact on quality of life). Maximum Score: 30 (extremely large impact on quality of life).

SECONDARY OUTCOMES:
Physician assessed body surface area affected | baseline, week 8 and 16
  Range from 0% (no affected area) to 100% (complete involvement)
Investigator/physician global assessment | baseline, week 8, week 16
  0 to 5 point numerical rating scale, with a higher value signalling greater severity
Eczema severity | baseline, week 8, week 16
  Eczema Area and Severity Index. Scoring system used to assess the severity of atopic dermatitis. Score ranges from 0 to 72 with higher score indicating worse severity.
Psoriasis Severity | baseline, week 8, week 16
  Psoriasis Area and Severity Index. Severity assessment for patients with psoriasis. Score ranges from 0-72 with higher scoring indicating more severe disease.
Chronic urticaria severity | baseline, week 8, week 16
  Urticaria Activity Score-7 (UAS7). Assess severity for patients with chronic urticaria. Score ranges from 0-6.
Composite measure of scratching | baseline, week 8, week 16
  Global severity and body surface area affected of various scratching measures e.g excoriation, lichenification, prurigo
Itch | baseline, weeks 4, 8, 12, 16, 24, 32
  0-10 numerical rating scale, with higher scores signalling greater itch
Skin pain | baseline, week 4, week 8, week 12, week 16, week 24, week 32
  0-10 numerical rating scale, greater scores signalling greater pain
Sleep disturbance | baseline, weeks 4, 8, 12, 16, 24, 32
  0-10 numerical rating scale, with higher scores signalling greater sleep disturbance
Depression | baseline, week 8, week 16, week 24 and 32
  PROMIS (Patient-Reported Outcomes Measurement Information System) Depression 8b. The raw score range for the PROMIS Depression 8b ranges from 8 to 40 with higher scores indicating greater depressive symptoms. The raw score is then converted to a T-score using a standardized conversion table. The T scores have a mean of 50 and standard deviation (SD) of 10, a higher value signals greater depressive symptoms.
Anxiety | baseline, weeks 8, 16, 24 and 32
  PROMIS (Patient-Reported Outcomes Measurement Information System) Anxiety 7a. The raw score range from 7-35 with higher scores indicating greater anxiety symptoms. The raw score is then converted to a T-score using a standardized conversion table. The T scores have a mean of 50 and standard deviation (SD) of 10, a higher value signals greater depressive symptoms.
Number of patients requiring treatment escalation | baseline, week 8, 16 and 32
  Number of patients requiring treatment escalation, defined as any of the following
  - Initiation or escalation of systemic treatments; inclusive of conventional immunosuppressants, biologics, systemic steroids
Work productivity and activity impairment | baseline and week 16
  Modified Work Productivity and Activity Impairment Questionnaire plus Classroom Impairment Questions: SHP, Version 2 (WPAI+CIQ:SHP, V 2). Assesses the impact of health problems on a person's ability to work and perform regular daily activities. Scores are multiplied by 100 to express in percentages with higher scorings indicating greater impairment and less productivity.
  Two additional questions assessing time spent on problems associated with skin condition and employment status, respectively.
EQ-5D-5L | baseline, week 32
  EuroQol Group EQ-5D is a measure of health state/health utility. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state
Skin-specific quality of life impairment | week 4, week 12, week 16, week 24, week 32
  Dermatology Life Quality Index (DLQI). Minimum Score: 0 (no impact on quality of life). Maximum Score: 30 (large impact on quality of life).
Implementability - App Engagement Scale | week 32
  App Engagement Scale. 7 questions graded on a likert scale. Items are summed, with scores ranging from 7 to 35, with a higher score indicating greater engagement.
Implementability - Frequency of app usage | week 8, week 32
  Frequency of using the mobile app, ranging from never to everyday
Implementability - Duration of app usage | week 8, week 32
  Average duration of app use each time, ranging from less than 2 minutes to more than 40 minutes.
Implementability - Willingness to pay | week 32
  Single bounded willingness to pay, 'How much would you maximally be willing to pay/month to continue using this mobile app?' with responses ranging from 'I would not use it even if free' to 'I would pay $41 or more /month'
Implementability - Barriers and facilitators of use | Post 32 weeks after participant's study completion
  Qualitative interviews with thematic analysis to determine barriers and facilitators of use and long term sustainability
Implementability - Percentage completed learning paths/ modules | baseline to week 32
  Passively collected in mobile app's logs.
Implementability - Appropriate responses and engagement to tracking exercises and open ended questions in the app | Baseline to week 32
  Passive collected in mobile app's logs.
Implementability - Collective server statistics | baseline to week 32
  Mobile app's collective server access statistics is tracked to determine which pages have the lowest and highest traffic and to analyse 'helpfulness' ratings of each module.
Implementability - Likely frequency of app use after study | week 32
  Likely frequency of app usage after the study, ranging from never to everyday.
Implementability - Likes and dislikes | week 32
  Two free-text questions collecting qualitative feedback on participants' likes and dislikes about the app, respectively.
Implementability - Suggestions and feedback | week 32
  Free-text question collecting suggestions and feedback to improve the mobile app.
Physician assessed global disease severity | baseline, week 8, week 16
  Assesses patient's overall, emotional, functional, and physical severity, and physician's perception of how the patient graded overall severity. Range from 0 to 10, with higher value signalling greater severity.
Physician assessed clinical global change | week 8, week 16
  Clinician-assessed change in patient's overall status since the start of the study. Ranges from very much improved to very much worse.
Patient's disease severity grading | baseline, week 4, week 8, week 12, week 16, week 24, week 32
  A question assessing patient's overall global assessment of disease severity, ranging from 0 to 10, with higher scores indicating higher severity.
Patient Global Impression of Severity | baseline, week 4, week 8, week 12, week 16, week 24, week 32
  Patient reported global severity rating, ranging from none to very severe.
Patient Global Impression of Change | week 4, week 8, week 12, week 16, week 24, week 32
  Patient reported change in overall status from the start of the study, ranging form very much improved to very much worse.

OTHER OUTCOMES:
Type D personality | baseline and week 16
  DS-14, measure of type D personality. The negative affect and social inhibition scales are scored from 0-28 with a higher score representing greater trait. A cutoff of 10 on each scale is used to classify type D personality.
Itch characteristic | 0, week 8
  5D Pruritus scale ranges from 5 to 25, where 5 indicates no pruritus and 25 indicates the most severe pruritus.
Scratching behavior | baseline, week 8, week 16, week 24, week 32
  PROMIS Itch Questionnaire Scratching Behaviour 5a. Score ranges fro 0-25 with higher score indicating greater scratching behaviours. Scores are standardized with 50 representing the mean.
Acceptance of health condition | baseline, week 8, week 16, 32
  Acceptance of Chronic Health Conditions Scale. Scores range from 8 to 40. Higher scores indicate greater acceptance of the chronic health condition.
Revised illness perception questionnaire | baseline, week 8, week 16, 32
  Assessment of how individuals perceive their illness including cognitive and emotional representations of illness across several dimensions. Each dimension is scored separately and expressed as a percentage (0-100%), with higher scores indicating more strongly held beliefs.
Resilience | baseline, week 8, week 16, 24, 32
  Brief Resilience Scale. The total score on the Brief Resilience Scale (BRS) ranges from 6 to 30. This scale measures an individual's ability to bounce back from stress and adversity. A higher score indicates greater resilience, while a lower score suggests lower resilience.
Self Efficacy in managing emotions | baseline, week 8, 32
  PROMIS self-efficacy in managing emotions 4a. Score ranges from 4 to 20 which are standardized and expressed as a percentage from 0-100%, with higher score indicating greater self efficacy.
Mindfulness | baseline, week 8, 32
  2 questions from the Cognitive and Affective Mindfulness Scale- Revised (CAMS-R). Score ranges from 0-6 with higher score indicating more mindfulness.
Self stigmatization | baseline, week 8, week 16, 32
  Weight bias internalization scale, modified for skin conditions. The score ranges from 11 to 77. Higher scores indicate greater internalization of bias/negative perception towards self.
Social Comparison | baseline, week 8, week 16, 32
  The DermSC scale comprises 3 questions, testing the general tendency for social comparison, downward negative comparison and upward negative comparison. The scores of each question (1-5 points) are tabulated (range 3-15) with a higher score indicating a greater degree of social comparison.
Well being | baseline, week 8, week 16, 24, 32
  World Health Organisation-Five Well-Being Index (WHO-5) ranges from 0-25 which is converted to an index score 0-100 with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Adherence | baseline, week 8, week 16, 32
  Self-reported treatment adherence, represented as a percentage from 0-100% where higher scores indicate greater adherence.
Self-efficacy for managing social interactions | baseline, week 8, week 32
  2 questions from PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Social Interactions. It assesses confidence in social activities and help seeking, ranging from I am not at confident to I am very confident.

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Choi, MBBS, Principal Investigator — National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Yes
IPD shared includes de-identified demographics, disease outcomes and measures.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD and supporting information will be available from the time of publication and for four years thereafter.
Access Criteria: IPD and supporting information will be available from the study team on a case-by-case basis upon request.

REFERENCES:
- [Derived] Choi E, Long V, Phan P, Shen L, Lim ZV, Koh MJ, Chua JY, Dalakoti M, Ho CS, Chandran NS, Sevdalis N, Valderas JM, Hsu KJ. Protocol for a double-blinded randomised controlled trial and process evaluation of a digital psychotherapeutic app in Singapore to improve symptom burden in patients with dermatological problems. BMJ Open. 2025 Jul 25;15(7):e098266. doi: 10.1136/bmjopen-2024-098266. PMID 40713034